CLINICAL TRIAL: NCT02698826
Title: Reoxygenation After Cardiac Arrest II (REOX II Study)
Acronym: REOX II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REOX II; R01HL112815 (NIH)
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest, Hyperoxia, Ischemia-reperfusion Injury, Reactive Oxygen Species, Oxidative Stress, Neuropsychological Tests
MeSH Terms: conditions — Heart Arrest; Hyperoxia; Reperfusion Injury | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adult patients resuscitated from cardiac arrest (Experimental): Rapid FiO2 optimization protocol
  Interventions: Other: Protocol for rapid FiO2 optimization

INTERVENTIONS:
Other: Protocol for rapid FiO2 optimization — We plan to test a protocol for FiO2 optimization for mechanically ventilated post-cardiac arrest subjects, with a therapeutic goal of partial pressure of arterial oxygen (PaO2) of 60-99 mmHg, based on the PaO2 range that was associated with the lowest risk of poor outcome in our previously published work. We also use PaO2 (measured by arterial blood gas [ABG] analysis) as the ultimate goal rather than arterial oxygen saturation (SaO2) measured by pulse oximetry because an SaO2 value <100% on pulse oximetry monitoring does not always exclude supranormal PaO2. The protocol in this application begins with very rapid reduction of FiO2 as much as possible according to SaO2 values, and when FiO2 is maximally reduced by SaO2 an ABG is measured, followed by finer adjustment of FiO2 to achieve a PaO2 60-99 mmHg. The protocol not only prescribes each downward titration of FiO2 but it also includes detailed limbs for upward titration of FiO2 to account for potential "overshoot" in FiO2 reduction.

SUMMARY:
The broad objective of this study is to test the association between hyperoxia exposure after resuscitation from cardiac arrest and outcome. After obtaining written informed consent subjects enrolled in REOX II will undergo a rapid faction of inspired oxygen (FiO2) optimization protocol to prevent exposure to hyperoxia. We will compare outcomes between subjects enrolled in REOX I (observational study only) and REOX II (intervention: rapid FiO2 optimization protocol). Our overarching hypothesis is that exposure to hyperoxia after return of spontaneous circulation (ROSC) is associated with increased oxidative stress and worsened neurological and cognitive outcomes.

DETAILED DESCRIPTION:
Specific Aim 1: Test if initiation of the rapid FiO2 optimization protocol following ROSC from cardiac arrest is associated with the degree of in vivo oxidative stress during the post-resuscitation phase of therapy.

Approach: We will conduct a multicenter interventional study (FiO2 optimization protocol) of adult patients resuscitated from cardiac arrest. We will record data pertaining to oxygenation parameters and other factors and measure biomarkers of oxidative stress [isoprostanes (IsoPs) and isofurans (IsoFs)] in the plasma at 0 and 6 hours after ROSC using gas chromatography negative ion chemical ionization mass spectrometry. We will compare plasma IsoPs/IsoFs at each time point between subjects enrolled in REOX II (i.e. receive the study intervention, rapid FiO2 optimization) and REOX I (i.e. do not receive the study intervention) using t-test or Mann-Whitney U as appropriate with corrections for multiple comparisons.

Specific Aim 2: Test if initiation of the rapid FiO2 optimization protocol following ROSC from cardiac arrest is associated with a decrease in neurological disability at hospital discharge.

Approach: In the study described above, we will determine the Modified Rankin Scale (mRS) at hospital discharge. We will compare proportions of good neurological outcome [defined as a mRS ≤ 3] between subjects enrolled in REOX II (i.e. receive the study intervention, rapid FiO2 optimization) vs. those enrolled in REOX I (i.e. do not receive the study intervention), using binomial test.

Specific Aim 3: Test if initiation of the rapid FiO2 optimization protocol following ROSC from cardiac arrest is associated with neuropsychological outcomes among survivors at 180 days.

Approach: In the study described above, we will assess neuropsychological outcome among survivors at 180 days. Neuropsychological testing will use validated instruments across five cognitive domains (attention, Wechsler Adult Intelligence Scale-IV-digit span; (2) reasoning, Wechsler Adult Intelligence Scale-IV-similarities; (3) immediate and delayed memory, Wechsler Memory Scale-III-logical memory I and II; (4) verbal fluency, Controlled Oral Word Association Test; and (5) executive functioning, Hayling Sentence Completion Test). Among survivors, we will compare the 180-day neuropsychological measures (composite z-scores for each cognitive domain) between the same two groups using t-test or Mann-Whitney U as appropriate with corrections for multiple comparisons. We will also compare the proportions of patients able to return to work between the two groups using binomial test

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* Cardiac arrest
* Return of spontaneous circulation
* Not following commands immediately after ROSC
* Endotracheal intubation
* Clinician intent to treat with therapeutic hypothermia (or absence of clinician intent to withhold therapeutic hypothermia)

Exclusion Criteria:

* Presumed etiology of arrest is trauma
* Presumed etiology of arrest is hemorrhage
* Presumed etiology of arrest is sepsis
* Permanent resident of nursing home or other long-term care facility
* Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate, e.g. end stage chronic illness with no reasonable expectation of survival to hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Trzeciak, MD, MPH, Study Director — The Cooper Health System
Locations (5):
- United States (5):
  - Indiana University/ Methodist Hospital, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - Hospital of the University of Pennsylvania and Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Patients Resuscitated From Cardiac Arrest
Started | 16
Completed | 2
Not Completed | 14
Not completed — Death | 13
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- FiO2 Titration Group: Rapid FiO2 optimization protocol Protocol for rapid FiO2 optimization: We plan to test a protocol for FiO2 optimization for mechanically ventilated post-cardiac arrest subjects, with a therapeutic goal of partial pressure of arterial oxygen (PaO2) of 60-99 mmHg, based on the PaO2 range that was associated with the lowest risk of poor outcome in our previously published work. We also use PaO2 (measured by arterial blood gas [ABG] analysis) as the ultimate goal rather than arterial oxygen saturation (SaO2) measured by pulse oximetry because an SaO2 value <100% on pulse oximetry monitoring does not always exclude supranormal PaO2. The protocol in this application begins with very rapid reduction of FiO2 as much as possible according to SaO2 values, and when FiO2 is maximally reduced by SaO2 an ABG is measured, followed by finer adjustment of FiO2 to achieve a PaO2 60-99 mmHg. The protocol not only prescribes each downward titration of FiO2 but it also includes detailed limbs for upward titration of FiO2 to account for potential "overshoot" in FiO2 reduction.
Arm/Group | FiO2 Titration Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Plasma Isofurans (pg/mL)/Isoprostanes (pg/mL) Ratio
Time Frame: Change in the isofurans/isoprostanes ratio between 0 and 6 hours post-ROSC
Population: Not analyzed secondary to no measurements obtained for intervention arm.
Groups:
- FiO2 Titration: Not analyzed secondary to insufficient samples
Arm/Group | FiO2 Titration
Number analyzed (Participants) | 0

2. Secondary Outcome: Modified Rankin Scale (mRS) (Primary Neurological Outcome)
Description: 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: Upon hospital discharge, on average two weeks
Measure: Median (Full Range); unit: score on a scale
Groups:
- FiO2 Titration: Single arm
Arm/Group | FiO2 Titration
Number analyzed (Participants) | 16
score on a scale | 6 [0 to 6]

3. Other Pre Specified Outcome: Composite Neuropsychological Testing Score
Description: The neuropsychological testing uses validated instruments across five cognitive domains: (1) attention, Wechsler Adult Intelligence Scale-IV-digit span; (2) reasoning, Wechsler Adult Intelligence Scale-IV-similarities; (3) immediate and delayed memory, Wechsler Memory Scale-III-logical memory I and II; (4) verbal fluency, Controlled Oral Word Association Test; and (5) executive functioning, Hayling Sentence Completion Test.
Time Frame: 180 days
Population: No analysis performed secondary to no patients were able to undergo the neuropsychological testing.
Groups:
- FiO2 Titration: Insufficient survivors to analyze.
Arm/Group | FiO2 Titration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | FiO2 Titration
All-Cause Mortality (participants affected / at risk) | 13/16
Serious Adverse Events (participants affected / at risk) | 14/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FiO2 Titration (N=16)
Death (Cardiac disorders) | 13 (13)
Poor neurological outcome (Nervous system disorders) | 1 (1) — Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance or Severe disability; bedridden, incontinent and requiring constant nursing care and attention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02698826/Prot_SAP_000.pdf